CLINICAL TRIAL: NCT07004062
Title: Application Value of Targeted Nursing Based on Risk Assessment Strategies in the Treatment of Patients With Gynecological Endocrine Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Obstetrics and Gynecology Hospital of Fudan University-Huangpu Campus (Other Government)
Responsible Party: Principal Investigator, Haiyan Wang, Principal Investigator, Obstetrics and Gynecology Hospital of Fudan University-Huangpu Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: No.20230815
Record Dates: First submitted 2025-05-15; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2023-12

CONDITIONS: Gynecological Endocrine Disorders; Risk Assessment; Targeted Nursing Care; Psychological Support; Quality of Life

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): In the control group, patients received routine nursing care, which primarily involved regular monitoring of vital signs such as blood pressure, temperature, pulse, and respiration. Basic health education was provided, focusing on lifestyle guidance including dietary control and daily routine recommendations. General psychological support was offered through emotional soothing and communicative care to alleviate anxiety. Medication management was strictly implemented in accordance with medical orders to ensure accurate drug administration. In addition, basic daily nursing operations were performed, including assistance with personal hygiene, regular turning to prevent pressure sores, and therapeutic massage when necessary.
  Interventions: Other: Structured Risk Assessment-Based Targeted Nursing Intervention
- observation group (Experimental): Patients in the observation group, on the other hand, received targeted nursing interventions based on a structured risk assessment strategy in addition to routine care. This included a comprehensive individualized health assessment that evaluated the patient's lifestyle, dietary habits, stress levels, sleep quality, medical history, and level of social support, leading to the formulation of a personalized nursing plan. Emotional and psychological support was intensified for patients experiencing emotional instability, employing interventions such as cognitive-behavioral therapy, relaxation training, and stress management techniques. Lifestyle interventions were also enhanced by guiding patients to establish regular routines, adopt low-sugar and high-fiber diets rich in vitamins, and engage in appropriate physical activity. Professional nursing interventions were applied to patients with menstrual irregularities or fertility-related needs, including ovulation monitoring and reproducti
  Interventions: Other: Structured Risk Assessment-Based Targeted Nursing Intervention

INTERVENTIONS:
Other: Structured Risk Assessment-Based Targeted Nursing Intervention — Comprehensive Risk Assessment: Evaluation of lifestyle factors (diet, exercise, sleep), psychosocial stressors, medical history, and endocrine-specific biomarkers
  Personalized Care Plan: Tailored interventions addressing identified risk factors
  Psychological Component: Cognitive-behavioral techniques and stress management
  Lifestyle Modification: Guided nutrition (low-glycemic, high-fiber diet) and physical activity plans
  Reproductive Health Support: Menstrual cycle monitoring and fertility-related counseling

SUMMARY:
Risk-based targeted nursing significantly enhances clinical outcomes, quality of life, and mental health in patients with gynecological endocrine disorders, supporting its broader clinical application.

DETAILED DESCRIPTION:
To evaluate the clinical value of targeted nursing care based on risk assessment in patients with gynecological endocrine disorders.

A prospective controlled study was conducted to analyze the clinical data of 84 patients with endocrine disorders and 89 healthy women, focusing on identifying risk factors associated with endocrine disorders and designing corresponding personalized nursing interventions. A total of 154 patients with gynecological endocrine disorders, treated between December 2023 and June 2024, were randomly assigned into a control group (n = 77) and an observation group (n = 77) using a random number table method. The control group received routine nursing care, while the observation group received targeted nursing interventions based on risk assessment strategies in addition to routine care. Nursing outcomes, patient satisfaction, quality of life scores, and psychological status-including Self-Rating Anxiety Scale (SAS) and Self-Rating Depression Scale (SDS) scores-were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of gynecological endocrine disorder

Aged 18-45 years

Complete clinical data available

Willing and able to provide informed consent

Exclusion Criteria:

Severe systemic or psychiatric illness

Recent major surgery or hormonal/fertility treatment (within 3 months)

Known hypersensitivity to study medications

Currently pregnant or breastfeeding

Participation in another clinical trial within 6 months

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Clinical Efficacy of Targeted Nursing in Gynecological Endocrine Disorders | Baseline to 6 months post-intervention.
  Proportion of patients achieving significant improvement in endocrine symptoms (e.g., menstrual regularity, hormonal balance) post-intervention, assessed via physician evaluation and laboratory markers (e.g., LH/FSH ratio, testosterone levels).

SECONDARY OUTCOMES:
Patient Satisfaction with Nursing Care | End of intervention (Week 12).
  Satisfaction rates measured via a 5-point Likert scale survey (1 = "very dissatisfied" to 5 = "very satisfied"), including domains of communication, pain management, and emotional support.

OTHER OUTCOMES:
Adherence to Lifestyle Interventions | Weekly during intervention (Weeks 1-12).
  Proportion of patients adhering to prescribed diet/exercise plans, recorded via self-reported logs and nurse audits.

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China